CLINICAL TRIAL: NCT02961218
Title: A Multiple-dose, Subject- and Investigator-blinded, Placebo-controlled, Parallel Design Study to Assess the Efficacy, Safety and Tolerability of ACZ885 (Canakinumab) in Pediatric and Young Adult Patients With Sickle Cell Anemia
Brief Title: Study of Efficacy, Safety and Tolerability of ACZ885 (Canakinumab) in Pediatric and Young Adult Patients With Sickle Cell Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885X2206
Record Dates: First submitted 2016-10-20; First posted 2016-11-10 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle cell disease; hemoglobinopathy; pediatric
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Monthly doses of 4 mg/kg for subjects weighing ≤40 kg and 300 mg for all other subjects
  Interventions: Drug: Placebo
- ACZ885 (Experimental): Monthly doses of 300 mg (4 mg/kg for patients ≤ 40 kg) canakinumab s.c.
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885 — Monthly doses of 4 mg/kg for subjects weighing ≤40 kg and 300 mg for all other subjects
  Other Names: Canakinumab
  Arms: ACZ885
Drug: Placebo — Monthly doses of placebo to match the administered dose of canakinumab s.c.
  Arms: Placebo

SUMMARY:
The study assesses the efficacy, safety and tolerability of ACZ885 (canakinumab) in pediatric and young adult patients with sickle cell anemia (SCA).

DETAILED DESCRIPTION:
This was an ambulatory-based 24-week study followed by an additional 24-week open label phase. It was a subject- and investigator-blinded, randomized, placebo-controlled, parallel group, non-confirmatory study to assess the clinical efficacy of ACZ885 administered s.c. in six injections given 28 days apart (in each phase of the study).

Pediatric and young adult subjects diagnosed with sickle cell anemia (SCA) were planned to be randomized to either ACZ885 treatment or placebo treatment in a 1:1 ratio,.

For each subject, there was a maximum 28-day screening period that included recording of daily pain frequency and intensity by e-diary for at least 1 week. Subjects who met the eligibility criteria at screening underwent evaluation of baseline clinical and biomarker assessments prior to first dose administration.

On Day 1, monthly s.c. dosing with ACZ885 started at 4 mg/kg for subjects weighing ≤40 kg and 300 mg for all other subjects. Subjects in the placebo treatment arm were injected with placebo in a like manner. All subjects returned to the study centers for safety checks on a monthly basis when they received treatment with either ACZ885 or placebo.

The final blinded dosing was given on Week 20, followed by blinded clinical assessments at Week 24. Subjects from both study arms were then offered optional, open label monthly dosing of ACZ885 for an additional 24 weeks (Weeks 24-48) with clinical outcome assessment.

Subjects returned for the end of study (EOS) visit at Week 56. For subjects who chose not to participate in the optional, open label portion of the study, or for those stopping treatment early for any other reason, an EOS visit occurred approximately 8 weeks after last dose received.

After enrollment of 49 subjects, Novartis decided to terminate the study early due to strategic reasons not related to safety and decided that no additional enrollment was needed in order to interpret the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 8-20 years of age (both inclusive) diagnosed with sickle cell anemia (HbSS) or sickle beta0 thalassemia (documented by family studies, or analysis of either hemoglobin or DNA).
* Patient's written informed consent from those ≥18 years of age must be obtained before any assessment is performed. Parent or legal guardian's written informed consent and child's assent, if appropriate, are required before any assessment is performed for patients < 18 years of age.
* Detectable baseline of background or episodic pain measured by daily e-diary over 1 to 2 weeks during screening period as defined below: Average daily pain score ≥ 1 cm without analgesic use over a period of at least 7 days and/or, At least one episode of pain requiring analgesic use during a period of up to 14 days.
* History of ≥2 vaso-occlusive pain episodes in the past year, as defined as pain with no other, non-sickle cell identifiable cause that requires analgesia and interferes with the patient's normal daily routine.

Exclusion Criteria:

* History of known hypersensitivity to canakinumab.
* Ongoing or treatment with the past 3 months with red blood cell transfusion therapy, or have evidence of iron overload requiring chelation therapy.
* Transcranial Doppler ultrasound in the past year or at screening in patients with an accessible transtemporal window, demonstrating velocity in middle or anterior cerebral or internal carotid artery ≥200 cm/sec.
* Administration of any other blood products within 3 weeks of screening visit.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Greenville, North Carolina
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Hamburg, Germany
- Novartis Investigative Site, Afula, Israel
- Novartis Investigative Site, Johannesburg, Guateng, South Africa
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Mersin
- United Kingdom (2):
  - Novartis Investigative Site, Wolverhampton, Staffordshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rees DC, Kilinc Y, Unal S, Dampier C, Pace BS, Kaya B, Trompeter S, Odame I, Mahlangu J, Unal S, Brent J, Grosse R, Fuh BR, Inusa BPD, Koren A, Leblebisatan G, Levin C, McNamara E, Meiser K, Hom D, Oliver SJ. A randomized, placebo-controlled, double-blind trial of canakinumab in children and young adults with sickle cell anemia. Blood. 2022 Apr 28;139(17):2642-2652. doi: 10.1182/blood.2021013674. PMID 35226723
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=849
- See also: A Pediatric Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 49 participants were randomized into the study from 15 centers in seven countries: Greater Britain (5), Israel (1), Germany (1), Turkey (3), South Africa (1), USA (3) and Canada (1).
Pre-assignment Details: Subjects who met the eligibility criteria at screening underwent evaluation of baseline clinical and biomarker assessments prior to first dose administration.
Groups:
- Placebo: Monthly doses of placebo to match the administered dose of ACZ885 s.c.
Period: Overall Study
Arm/Group | ACZ885 | Placebo
Started | 25 | 24
Safety Analysis Set (included all subjects that received any study drug) | 25 | 24
Pharmacokinetics (PK) Analysis Set (included all subjects with at least one available valid PK concentration measurement) | 25 | 0 (Placebo patients were excluded from the PK analyses)
Primary PD Analysis Set (included all subjects with available PD data, who received any study drug.) | 25 | 24
Completed | 22 | 19
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Subject/Guardian Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACZ885 | Placebo | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.8 (2.69) | 15.6 (3.28) | 15.7 (2.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 12 | 13 | 25
  White | 12 | 10 | 22
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of 4- Week Average Daily Pain Measured by Visual Analog Score (VAS) Over the Period of Week 8 to 12
Description: Visual analog scale (VAS) was used to record severity. Pediatric and young adult participants rated their daily sickle cell associated pain intensity once each day in the evening using an 11-point numerical rating scale from 0 to 10 with higher ratings associated with more intense pain (0 = no pain, 10 = worst pain). For each subject, there was a maximum 28-day screening period that included recording of daily pain intensity by e-diary for at least 1 week. The average daily pain results in the screening period were used to derive the baseline value. The average over week 8 to 12 was calculated and the change from baseline in the average daily pain VAS was analyzed using a Bayesian model for repeated measures.
Time Frame: Baseline (upto 28 days prior to start of treatment), Week 8 to 12
Population: Pharmacodynamics (PD) analysis set: included all subjects with available PD data, who received any study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 25 | 24
Score on a scale | -0.45 (0.384) | -0.37 (0.402)
Statistical Analysis 1: Comparison: ACZ885 vs Placebo; Test type: Superiority; p = 0.55, Bayesian model for repeated measures — probability reduction of average pain score in ACZ885 > Placebo; Mean Difference (Net) = -0.07, 90% CI 2-sided [-1.03 to 0.85], Standard Deviation 0.57 — Lower limit and upper limit represents the credibility interval from the Bayesian analysis

2. Secondary Outcome: Change From Baseline of Average Daily Pain VAS Over 4 Weeks Intervals up to Week 24
Description: Visual analog scale (VAS) was used to record severity. Pediatric and young adult participants rated their daily sickle cell associated pain intensity once each day in the evening using an 11-point numerical rating scale from 0 to 10 with higher ratings associated with more intense pain (0 = no pain, 10 = worst pain). The average of 4 weeks interval up to week 24 was calculated.
Time Frame: Baseline (upto 28 days prior to start of treatment), Week 0 to 4, Week 4 to 8, Week 8 to 12, Week 12 to 16, Week 16 to 20 and Week 20 to 24
Population: Pharmacodynamics (PD) analysis set: included all subjects with available PD data, who received any study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 25 | 24
Score on a scale
  0-4 Weeks: number analyzed (Participants) | 25 | 23
  0-4 Weeks | -0.337 (1.629) | 0.007 (1.428)
  4-8 Weeks: number analyzed (Participants) | 22 | 20
  4-8 Weeks | -0.173 (1.515) | 0.158 (1.847)
  8-12 Weeks: number analyzed (Participants) | 21 | 18
  8-12 Weeks | -0.444 (1.437) | -0.376 (2.104)
  12-16 Weeks: number analyzed (Participants) | 19 | 20
  12-16 Weeks | -0.505 (1.744) | 0.057 (2.371)
  16-20 Weeks: number analyzed (Participants) | 25 | 16
  16-20 Weeks | -0.388 (1.772) | 0.151 (1.811)
  20-24 Weeks: number analyzed (Participants) | 17 | 16
  20-24 Weeks | -0.752 (1.678) | 0.036 (2.131)

3. Secondary Outcome: Change in the Concentration of High Sensitivity C-Reactive Protein (hsCRP) From Baseline to Week 12
Description: hs-CRP is a biomarker that represents the inflammation process.
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: mg/L
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 19
mg/L | 0.338 [0.237 to 0.483] | 0.830 [0.576 to 1.194]
Statistical Analysis 1: Comparison: ACZ885 vs Placebo; Test type: Superiority; p = 0.002, Mixed-effect Model for Repeated Measures; Ratio = 0.408, 90% CI 2-sided [0.253 to 0.658]

4. Secondary Outcome: Change in the Concentration of White Blood Cell (WBC) Count From Baseline to Week 12
Description: WBC count was used as a laboratory marker to determine the effect of the drug
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 19 | 17
10^9 cells/liter | 0.813 [0.737 to 0.898] | 1.081 [0.973 to 1.201]
Statistical Analysis 1: Comparison: ACZ885 vs Placebo; Test type: Superiority; p < .001, Mixed-effect Model for Repeated Measures; Ratio = 0.752, 90% CI 2-sided [0.657 to 0.862]

5. Secondary Outcome: Change in the Concentration of Absolute Count of Neutrophils From Baseline to Week 12
Description: Absolute count of neutrophils was measured as a laboratory marker to determine the effect of the drug
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 19 | 17
10^9 cells/liter | 0.717 [0.611 to 0.842] | 1.052 [0.888 to 1.246]
Statistical Analysis 1: Comparison: ACZ885 vs Placebo; Test type: Superiority; p = 0.004, Mixed-effect Model for Repeated Measures; Ratio = 0.682, 90% CI 2-sided [0.547 to 0.849]

6. Secondary Outcome: Change in the Concentration of Absolute Count of Blood Monocytes From Baseline to Week 12
Description: Absolute count of blood monocytes was measured as a laboratory marker to determine the effect of the drug.
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 19 | 17
10^9 cells/liter | 0.712 [0.590 to 0.859] | 0.992 [0.813 to 1.209]
Statistical Analysis 1: Comparison: ACZ885 vs Placebo; Test type: Superiority; p = 0.032, Mixed-effect Model for Repeated Measures; Ratio = 0.718, 90% CI 2-sided [0.556 to 0.925]

7. Secondary Outcome: Change in the Concentration of Hemoglobin From Baseline to Week 12
Description: Hemoglobin was used as a hemolysis marker to determine the effect of the drug.
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 19 | 19
g/L | -0.97 (4.727) | 1.11 (7.975)

8. Secondary Outcome: Change in the Reticulocyte Count From Baseline to Week 12
Description: Reticulocyte count was used as a hemolysis marker to determine the effect of the drug
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 18 | 19
10^9 cells/liter | -6.578 (64.1131) | 25.358 (47.6483)

9. Secondary Outcome: Change in the Concentration of Bilirubin From Baseline to Week 12
Description: Bilirubin was used as a hemolysis marker to determine the effect of the drug
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 19
umol/L | 5.05 (19.796) | -1.95 (11.591)

10. Secondary Outcome: Change in the Concentration of Lactate Dehydrogenase (LDH) From Baseline to Week 12
Description: LDH was used as a hemolysis marker to determine the effect of the drug
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 18 | 19
Units per liter (U/L) | 19.06 (70.862) | -33.74 (209.259)

11. Secondary Outcome: Change in the Concentration of Haptoglobin From Baseline to Week 12
Description: Haptoglobin was used as a hemolysis marker to determine the effect of the drug
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 13 | 19
g/L | -0.0112 (0.04022) | -0.0213 (0.07923)

12. Secondary Outcome: Change in the Concentration of Oxygen Percent Saturation (SAO2) From Baseline to Week 12
Description: SAO2 was used as a hemolysis marker to determine the effect of the drug
Time Frame: Baseline, Week 12
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Mean (Standard Deviation); unit: Oxygen Saturation Percent
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 20 | 19
Oxygen Saturation Percent | -0.5 (2.16) | -0.3 (1.82)

13. Secondary Outcome: Number of Days Absent From School or Work Due to Pain as Recorded by E-diary
Description: The number of SCA-related days absent from school or work were derived from eDiary records.
Time Frame: up to Week 24
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Mean (90% Confidence Interval); unit: Days
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 22 | 19
Days | 2.20 [1.69 to 2.70] | 1.86 [1.31 to 2.41]
Statistical Analysis 1: Comparison: ACZ885 vs Placebo; Test type: Superiority; p = 0.455, Generalized Linear Model (GLM); Ratio = 1.40, 90% CI 2-sided [0.58 to 3.40], Standard Error of Mean 0.45

14. Secondary Outcome: Number of Acute Blood Transfusions Per Patient by Study Period - Double-blind Period
Description: The occurrence of acute blood transfusions was summarized as the proportion of subjects who received at least one acute blood transfusion and the event rate of acute blood transfusions per subject, by study period, group and reason of transfusion.
Time Frame: 12 weeks
Population: Pharmacodynamics (PD) analysis including patients with a valid measurements for the outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 25 | 24
Participants
  Overall Acute blood transfusion: 0 transfusions | 20 | 18
  Overall Acute blood transfusion: 1 transfusion | 4 | 4
  Overall Acute blood transfusion: 2 transfusions | 1 | 1
  Overall Acute blood transfusion: 3 transfusions | 0 | 1
  Acute blood transfusion: Rescue: 0 transfusions | 23 | 19
  Acute blood transfusion: Rescue: 1 transfusion | 2 | 4
  Acute blood transfusion: Rescue: 2 transfusions | 0 | 1
  Acute blood transfusion: Rescue: 3 transfusions | 0 | 0
  Acute blood transfusion: Prophylactic: 0 transfusions | 22 | 22
  Acute blood transfusion: Prophylactic: 1 transfusion | 2 | 1
  Acute blood transfusion: Prophylactic: 2 transfusions | 1 | 1
  Acute blood transfusion: Prophylactic: 3 transfusions | 0 | 0

15. Secondary Outcome: Mean Serum Concentration After Repeated Dosing of ACZ885
Description: PK samples were collected at Baseline, Week 4, 12, 20 and 24. Mean and standard deviation of the ACZ885 concentration was reported. Only those participants available at the specified time points were analyzed
Time Frame: Baseline, Week 4, 12, 20 and 24
Population: Pharmacokinetics (PK) analysis set consisted of ACZ885 treated patients. Placebo patients were excluded from the PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACZ885
Number analyzed (Participants) | 25
ng/mL
  Baseline | 0 (0)
  Week 4: number analyzed (Participants) | 23
  Week 4 | 13100 (5490)
  Week 12: number analyzed (Participants) | 19
  Week 12 | 18700 (5860)
  Week 20: number analyzed (Participants) | 17
  Week 20 | 19700 (5810)
  Week 24: number analyzed (Participants) | 17
  Week 24 | 20600 (5930)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment (Week 48) plus 8 weeks post treatment, up to maximum duration of 56 weeks.
Description: Any sign or symptom collected in the double-blinded period i.e 24 weeks followed by an additional 24-week open label phase (optional). Adverse events were reported separately for the double-blind and the open-label phase.
Groups:
- ACZ885: Double-blind period (Week 0 to 24): Monthly doses of 4 mg/kg for subjects weighing ≤40 kg and 300 mg for all other subjects
- Placebo: Double-blind period (Week 0 to 24): Monthly doses of placebo to match the administered dose of ACZ885 s.c.
- ACZ885 / ACZ885: Open label Phase (after Week 24 to Week 56) for the participants originally randomized to ACZ885: Monthly doses of 4 mg/kg for subjects weighing ≤40 kg and 300 mg for all other subjects
- Placebo / ACZ885: Open label Phase (after Week 24 to Week 56) for the participants originally randomized to placebo: Monthly doses of 4 mg/kg for subjects weighing ≤40 kg and 300 mg for all other subjects
Arm/Group | ACZ885 | Placebo | ACZ885 / ACZ885 | Placebo / ACZ885
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 11/25 | 15/24 | 11/22 | 11/20
Other Adverse Events (participants affected / at risk) | 19/25 | 20/24 | 17/22 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 (N=25) | Placebo (N=24) | ACZ885 / ACZ885 (N=22) | Placebo / ACZ885 (N=20)
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 10 | 11 | 9 | 10
Asthenia (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Alloimmunisation (Immune system disorders) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 (N=25) | Placebo (N=24) | ACZ885 / ACZ885 (N=22) | Placebo / ACZ885 (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0
Medical device site irritation (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 3 | 2
Pain (General disorders) | 6 | 5 | 3 | 7
Pyrexia (General disorders) | 2 | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1 | 0
Allergy to metals (Immune system disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 2 | 6
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Oxygen saturation abnormal (Investigations) | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Spleen palpable (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Ultrasound Doppler abnormal (Investigations) | 0 | 1 | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 1 | 2 | 0 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 5
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Benign enlargement of the subarachnoid spaces (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 5 | 3 | 2 | 4
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Illness anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Pica (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 1
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Priapism (Reproductive system and breast disorders) | 0 | 2 | 0 | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT02961218/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02961218/SAP_000.pdf